CLINICAL TRIAL: NCT05823363
Title: Vaginal Cuff Infiltration With Liposomal Bupivacaine for Pain Relief: A Double Blind, Randomized Controlled Trial
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Maimonides Medical Center (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 2022-02-12
Record Dates: First submitted 2023-04-10; First posted 2023-04-21 (Actual); Last update posted 2025-03-19 (Actual); Status verified 2025-03

CONDITIONS: Postoperative Pain
Keywords: pain; bupivicaine; local infiltration
MeSH Terms: conditions — Pain, Postoperative; Pain

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Masking Description: double blind
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (2):
- Exparel and Bupivacaine Group (Experimental): The participants in this group will receive 10 ml of xxparel and 10 ml of bupivacaine in the vaginal cuff
  Interventions: Drug: Exparel with Bubivacaine
- Bupivacaine Only Group (Active Comparator): This group will receive 20ml of bupivicaine in the vaginal cuff
  Interventions: Drug: Bupivacaine only

INTERVENTIONS:
Drug: Exparel with Bubivacaine — 10ml Exparel mixed with10ml bupivicaine in vaginal cuff
  Arms: Exparel and Bupivacaine Group
Drug: Bupivacaine only — 20ml of Bubivacaine in the vaginal cugg
  Arms: Bupivacaine Only Group

SUMMARY:
The goal is to find out if Exparel (liposomal bupivacaine) given as an injection decreases pain score if given into the vaginal cuff right before starting the minimally invasive (robotic-assisted or laparoscopic) total hysterectomy in patients scheduled for benign indication? Participants will write down

1. pain score at various intervals
2. pain medication used Treatment patients will receive

1)intervention arm will receive Exparel mixed with bupivicaine 2)control arm will receive bupivicaine only

DETAILED DESCRIPTION:
The question is whether Exparel (liposomal bupivacaine) given as an injection decreases pain score if given into the vaginal cuff right before starting the minimally invasive (robotic-assisted or laparoscopic) total hysterectomy? A reduction in pain after the surgery would result in decrease in opioid usage, fewer opioid-related adverse events, and increased satisfaction in patients.

Intervention arm (40) will get 10ml of Exparel diluted with 10 ml of bupivacaine around 2,4, 8 and 10 o' clock in vaginal cuff. Placebo group (40) will receive 20 ml of normal saline in vaginal cuff. All women 35-75 years age range scheduled for Laparoscopic and robotic hysterectomies with Bilateral salpingectomy or bilateral salpingo-oophorectomy will be assessed for eligibility.

It is a prospective interventional study that involves use of liposomal bupivacaine and this study will be run in Maimonides medical center's gynecology department .

The severity of pain will be assessed preoperatively in the holding area, at the time of PACU arrival, and at 1hour, 12, 24, 48 and 72hours postoperatively using a VAS from 0 to 10 with 10 being the worst pain the patient has ever experienced. The first 3 assessments will be performed in the hospital by the principal investigators and the remaining assessments will happen through a phone conversation with the patient after discharge from hospital. The VAS has been found to be a simple scale.

The data will also be collected through chart review and. this data will include age, VAS score reporting by nurses in PACU, BMI, previous abdominal surgery, previous vaginal delivery and parity.

Pain inquiries will assess low pelvic/suprapubic area and lower abdominal pain, type of pain (dull, achy, sharp, stabbing, etc.) and radiation of pain to a surrounding area. Other endpoints will include number of patients who required break through (additional) opioid analgesic medications, median time to first break through opioid use, total opioid analgesic requirement. The time, day and number of requests for break-through (additional) analgesia will be noted by gynecologic surgery team (Research assistant) participating in this study.

When the patient is home the patient will have a Pain Medication Diary that the investigators will provide for the patient prior to discharge. Patient will be contacted over phone to get the data from her log sheet.

ELIGIBILITY:
Inclusion Criteria:

* Any patient age > 18 years who is having minimally invasive robotic or laparoscopic total hysterectomy for any indication without any anesthetic block.

Exclusion Criteria:

* 1) Use of any of the following medications within the times specified before surgery: a. opioid, SSRI, tricyclic antidepressant, gabapentin, pregabalin within three days of surgery. b. Use of acetaminophen within 24 hours of surgery 2) Concurrent painful physical condition or concurrent surgery that may require analgesic treatment (such as NSAID, opioid, SSRI, tricyclic antidepressant, gabapentin, pregabalin) in the postoperative period for pain that is not strictly related to the minimally invasive supracervical hysterectomy procedure and may confound the postoperative assessments (e.g., rheumatoid arthritis, chronic neuropathic pain.

  3) Chronic user of analgesic medications, including taking opioid medications for more than 14 days in the last 3 months, or nonopioid pain medications more than 5 times per week.

  4) Current use of systemic glucocorticosteroids (e.g. Decadron) or use of glucocorticoids within one month of enrollment into this study.

  5) History of hepatitis (other than hepatitis A). 6) History of hypersensitivity or idiosyncratic reactions to amide type local anesthetics, opioids, or propofol.

  7) Administration of an investigational drug within 30 days prior to study drug administration, or planned administration of another investigational product or procedure during the subject's participation in this study.

  8) Uncontrolled anxiety, schizophrenia, or other psychiatric disorder that, in the opinion of the Investigator, may interfere with study assessments or compliance.

  9) Significant medical conditions or laboratory results that, in the opinion of the Investigator indicate an increased vulnerability to study drug and procedures, and expose subjects to an unreasonable risk as a result of participating in this clinical trial.

  10) Any clinically significant event or condition uncovered during the surgery (e.g., excessive bleeding, acute sepsis) that might render the subject medically unstable or complicate the subject's postoperative course. 11) women with endometriosis 12) contraindications to any medication used in the study (acetaminophen, NSAID or opioid).

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 15 (Actual)
Dates: Start 2024-09-09 (Actual); Primary Completion 2024-09-09 (Actual); Study Completion 2024-09-09 (Actual)

PRIMARY OUTCOMES:
Pain reduction after surgery | 72 hours after surgery
  A reduction in pain on a 11 point Likert Scale with 0 being no pain and 10 being very severe pain.

CONTACTS AND LOCATIONS:
Overall Officials: Scott Chudnoff, MD, Principal Investigator — MMC
Locations (1):
- Maimonides Medical Center, Brooklyn, New York, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Ishio J, Komasawa N, Kido H, Minami T. Evaluation of ultrasound-guided posterior quadratus lumborum block for postoperative analgesia after laparoscopic gynecologic surgery. J Clin Anesth. 2017 Sep;41:1-4. doi: 10.1016/j.jclinane.2017.05.015. Epub 2017 Jun 1. PMID 28802593

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2022-12-29): https://cdn.clinicaltrials.gov/large-docs/63/NCT05823363/Prot_SAP_000.pdf